CLINICAL TRIAL: NCT01455610
Title: Preoperative Evaluation of Resectability of Pancreatic Head Cancer by Contrast-enhanced MDCT:a Multi-center Study
Brief Title: Resectability of Pancreatic Head Cancer by Contrast-enhanced MDCT:a Multi-center Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meng Su Zeng (Other)
Collaborators: Changhai Hospital (Other); Shanghai Cancer Hospital, China (Other); Ruijin Hospital (Other); Huashan Hospital (Other); Huadong Hospital (Other)
Responsible Party: Sponsor-Investigator, Meng Su Zeng, Mengsu Zeng, MD & Ph.D,Chairman & Professor,Department of Radiology, Shanghai Zhongshan Hospital
Organization: Shanghai Zhongshan Hospital (Other)
Other Study IDs: ZMS-001
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Adenocarcinoma of Head of Pancreas
Keywords: Computed tomography; Contrast enhancement; Pancreas; Cancer; Resectability
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this multicenter and double-blind clinical trial is to prospectively assess the sensitivity, specificity, negative predictive value, positive predictive value, and accuracy in respectability of pancreatic head cancer with contrasted-enhanced MDCT and its various post processing techniques, taking operational and pathological records as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients with (or suspected) pancreatic head cancer
* Being examined by contrasted-enhanced MDCT
* Receiving surgical treatment (including palliative surgery) in all research centers

Exclusion Criteria:

* Patients having (or suspected) pregnancy or breast-feeding
* Patients having allergic reactions to iodinated contrast agents or Hypersensitivity reactions to allergens(including drugs)
* Patients receiving ERCP before contrasted-enhanced MDCT examination
* Patients without surgery because of a high degree of surgical risk

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Out-patients or in-patients,with(or suspected) pancreatic head cancer, both have MDCT examinaton and receive surgery treatment
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2012-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mengsu Zeng, MD, PhD, Study Chair — Radiology Department, Zhongshan Hospital of Fudan University; Jianping Lu, MD,PhD, Principal Investigator — Radiology Department, Changhai Hospital Affiliated to Second Military Medical University; Weijun Peng, MD, PhD, Principal Investigator — Radiology Department, Cancer Hospital Affiliated to Fudan University; Fuhua Yan, MD, PhD, Principal Investigator — Radiology Department, Ruijin Hospital Affiliated to Shanghai Jiaotong University, China; Xiaoyuan Feng, MD, PhD, Principal Investigator — Radiology Department, Huashan Hospital, Fudan University, China; Yanqing Hua, MD, PhD, Principal Investigator — Radiology Department, Huadong Hospital Affiliated to Fudan University, China
Locations (6):
- China (6):
  - Radiology Department, Ruijing Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Radiology Department, Cancer Hospital, Fuandan University, Shanghai, Shanghai Municipality
  - Radiology Department, Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Radiology Department, Huadong Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Radiology Department, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Radiology Department, Changhai Hospital Affiliated to the Second Military Medical University, Shanghai, Shanghai Municipality